CLINICAL TRIAL: NCT05420363
Title: Influence of Surface Characteristics of Gait Training on Gait Kinematics and Walking Capacity in Children With Diplegic Cerebral Palsy
Brief Title: Influence of Surface Characteristics of Gait Training on Gait Kinematics and Walking Capacity in Children With Diplegic CP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shimaa Aly Mohamed saied, principle investigator, Cairo University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003599
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Diplegic Cerebral Palsy
Keywords: CP , Diplegia
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional physical therapy + gait training on different surfaces. (Experimental): Children in study group will receive designed physical therapy program in addition to gait training on different surfaces.
  Interventions: Other: different walking surfaces
- traditional physical therapy + traditional gait training (Experimental): -Children in control group will receive designed physical therapy program in addition to traditional gait training hard surface .
  Interventions: Other: traditional gait training over hard surface only

INTERVENTIONS:
Other: different walking surfaces — different surfaces materials and textures as sand ,grass, air mattress , foam mattress ,gravels and Rollator
  Arms: traditional physical therapy + gait training on different surfaces.
Other: traditional gait training over hard surface only — The children will receive gait training over hard surface and even ground only and bare feet without wearing any foot ware or orthosis
  Arms: traditional physical therapy + traditional gait training

SUMMARY:
Using challenging surfaces of gait training, which require constant adjustments of the body's movement patterns to maintain stability and provide different sensory and proprioceptive inputs to mimic real life situation is appropriate for children with CP. So, the purpose of the current study is to investigate the influence of surface characteristics of gait training on gait kinematics and walking capacity in children with diplegic CP.

DETAILED DESCRIPTION:
The purpose of the study is to determine the influence of surface characteristics (different surfaces materials and textures) of gait training on kinematics gait parameters (step length, step width, double support time and cadence) and the functional walking capacity in children with diplegic CP.

ELIGIBILITY:
Inclusion Criteria:

1. Their ages will range from 6 to 8 years old.
2. The degree of spasticity will range from grade 1 or 1+ according to Modified Ashworth Scale.
3. They will be at level II on GMFCS .
4. They will be able to follow verbal command or instructions.

Exclusion Criteria:

* 1. Fixed deformities of lower limbs. 2. Sever visual or auditory problems. 3. History of surgical interference in lower limbs less than one year. 4. Botulinum toxin injections to the lower limb during the previous 4 months.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
kinematics gait parameters | over 3 months
  step length
kinematics gait parameters | over 3 months
  step width
kinematics gait parameters | over 3 months
  double support time
kinematics gait parameters | over 3 months
  cadence

SECONDARY OUTCOMES:
Six-minute walking test | over 3 months
  The 6-minute walk test (6MWT) is self-paced walking test commonly used to assess functional capacity in children with CP. It can be easily applied in clinical sitting; it reflects functional capacity in terms of activities of daily living

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university , Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No